CLINICAL TRIAL: NCT02152358
Title: Efficacy of a Preemptive Treatment by Ganciclovir or by Aciclovir in ICU Patients Requiring Prolonged Mechanical Ventilation and Presenting a Viral Replication (CMV and/or HSV) - Prospective, Randomized, Double-blinded Multicenter Trial
Brief Title: PTH - Preemptive Treatment for Herpesviridae
Acronym: PTH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20126003312-30; 2012-003312-30 (EudraCT Number)
Record Dates: First submitted 2014-03-26; First posted 2014-06-02 (Estimated); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Viral Pneumonia
Keywords: Cytomegalovirus; Herpes simplex virus; ICU; mechanical ventilation; mortality; ventilator-free days; PCR
MeSH Terms: conditions — Pneumonia, Viral; Herpes Simplex | interventions — Acyclovir; Ganciclovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Ganciclovir (Active Comparator): Patients with a positive CMV PCR
  Interventions: Drug: Ganciclovir
- Ganciclovir placebo (Placebo Comparator): Patients with a positive CMV PCR
  Interventions: Drug: Placebo
- Aciclovir (Active Comparator): Patients with a PCR positive for HSV
  Interventions: Drug: Aciclovir
- Aciclovir placebo (Placebo Comparator): Patients with a positive PCR for HSV
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aciclovir — Intravenous 15 mg/kg/d during 14 days
  Arms: Aciclovir
Drug: Ganciclovir — intravenous 10 mg/kg/d for 14 days
  Arms: Ganciclovir
Drug: Placebo
  Arms: Aciclovir placebo; Ganciclovir placebo

SUMMARY:
The aim of this study is to show that a preemptive treatment by ganciclovir (for positive CMV viremia) or aciclovir (for positive HSV oro-pharyngeal PCR) is able to increase the number of ventilator-free days at Day 60.

ELIGIBILITY:
Inclusion Criteria:

* mechanical ventilation > 96 hrs and expected duration of mechanical ventilation of at least 2 days
* positive blood CMV PCR (500 IU/ml) OR positive oropharyngeal HSV PCR
* age > 18 years
* informed consent
* negative pregnancy test

Exclusion Criteria:

* < 18 years
* Receiving ganciclovir or aciclovir or another antiviral agent active against HSV/CMV
* Had received antiviral agent active against HSV/CMV during the previous month
* Hypersensitivity to aciclovir/ganciclovir
* Pregnancy
* Breast feeding
* Bone marrow failure
* Solid organ recipients
* Bone marrow recipients
* HIV positive patients
* Receiving immunosuppressive agents
* SAPS II > 75
* Withdrawing/withholding
* Neutropenia (< 500 mm3)
* Thrombocytopenia (< 25 G/L)
* ICU readmission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2014-02-05 (Actual); Primary Completion 2018-04-21 (Actual); Study Completion 2023-04-05 (Actual)

PRIMARY OUTCOMES:
Ventilator-free days at Day 60 | 60 days

SECONDARY OUTCOMES:
Day 60 mortality | 60 days
ICU mortality | 60 days
Hospital mortality | 60 days
Duration of mechanical ventilation in survivors | 60 days
Duration of ICU stay | 60 days
Duration of hospital stay | 60 days
Incidence of ventilator-associated pneumonia | 60 days
Incidence of bacteremia | 60 days
SOFA score | days 3, 5, 7, 14, 21 and 28
Acute renal failure related to aciclovir or its placebo | 60 days
Leucopenia related to ganciclovir or its placebo | 60 days
Time to oropharyngeal negativation of HSV PCR | 30 days
Time to blood negativation of CMV PCR | 30 days
Incidence of herpetic bronchopneumonia | 60 days
Incidence of active CMV infection | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Papazian, MD, PhD, Principal Investigator — APHM - AMU
Locations (1):
- Assistance Publique - Hôpitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Luyt CE, Forel JM, Hajage D, Jaber S, Cayot-Constantin S, Rimmele T, Coupez E, Lu Q, Diallo MH, Penot-Ragon C, Clavel M, Schwebel C, Timsit JF, Bedos JP, Hauw-Berlemont C, Bourenne J, Mayaux J, Lefrant JY, Mira JP, Combes A, Wolff M, Chastre J, Papazian L; Preemptive Treatment for Herpesviridae Study Group, Reseau Europeen de recherche en Ventilation Artificielle Network. Acyclovir for Mechanically Ventilated Patients With Herpes Simplex Virus Oropharyngeal Reactivation: A Randomized Clinical Trial. JAMA Intern Med. 2020 Feb 1;180(2):263-272. doi: 10.1001/jamainternmed.2019.5713. PMID 31841577